CLINICAL TRIAL: NCT05630703
Title: Trial of Mindfulness-based Irritable Bowel Syndrome Eating Awareness Training as Compared to the Standard Low Fermentable Oligosaccharide, Disaccharide, Monosaccharide and Polyol Diet in Patients With Irritable Bowel Syndrome (IBS)
Brief Title: Mindfulness Training Versus Low (FODMAP) Fermentable Oligosaccharides, Disaccharides, Monosaccharides and Polyols Diet
Acronym: FODMAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00083217; 07-19-15E (Other: Atrium Health)
Record Dates: First submitted 2022-11-15; First posted 2022-11-30 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-08

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Irritable Bowel Syndrome (IBS); Mindfulness; FODMAP
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet; Diet Therapy

STUDY DESIGN:
Intervention Model Description: The randomization scheme used will be a random number generator using the Research Randomizer website (https://www.randomizer.org/) where the subjects will be randomized in one (1) of two (2) arms:
  Mindfulness-based Awareness Training in IBS (MB-IBS-EAT) Intervention OR Low FODMAP Diet Intervention
Who Masked: Investigator
Masking Description: The principal investigator will be blinded for the duration of the study. The study psychologist and the dietician will be blinded to the study results for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Training (Experimental): Behavioral: Mindfulness-based Eating Awareness Training in IBS - The MB-IBS-EAT is an 8-week intervention with weekly 1-hour sessions in a web-based group format.
  Interventions: Behavioral: Mindfulness-based Attention Training in IBS
- fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAP) diet (Active Comparator): Dietary: Low FODMAP Diet - Subjects in the FODMAP group will be provided dietary instructions by a registered dietician during weekly 1-hour sessions in a web-based group format.
  Interventions: Other: Low FODMAP Diet

INTERVENTIONS:
Behavioral: Mindfulness-based Attention Training in IBS — The MB-IBS-EAT is an 8-week intervention with weekly 1-hour sessions in a web-based group format.
  Arms: Mindfulness Training
Other: Low FODMAP Diet — Subjects in the FODMAP group will be provided dietary instructions by a registered dietician during weekly 1-hour sessions in a web-based group format
  Other Names: Dietary Intervention
  Arms: fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAP) diet

SUMMARY:
The study aims to compare the effect of mindfulness-based awareness training in Irritable Bowel Syndrome (IBS) (MB-IBS-EAT) with the dietary standard of care (low fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAP) diet) on patient's IBS symptoms

DETAILED DESCRIPTION:
This pilot study will be a randomized parallel trial comparing MB-IBS-EAT done over an 8-week period to a standard low FODMAP diet. The low FODMAP diet is currently employed by clinicians as a treatment for IBS, but response rates are poor, without documented long-term benefit. This finding supports the need for better, longer lasting interventions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Meets Rome IV criteria for diagnosis of Irritable Bowel Syndrome (IBS)
* Has legal and mental capacity to understand and sign an informed consent document
* Access to a computer or smart device with internet

Exclusion Criteria:

* Pregnancy
* Active malignancy in the previous five years
* Current or prior history of alcohol or drug abuse as defined by clinician
* Any history of eating disorder such as anorexia or bulimia
* Taking yoga or with prior history of mindfulness therapy within 3 months of enrollment
* Currently on a fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAP) diet
* Psychiatric illnesses other than depression or anxiety disorder
* Nausea or vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Global Improvement Scale (GIS) Scores Baseline | Baseline
  The Global Improvement Scale is an overall assessment of Irritable Bowel Syndrome (IBS) symptoms using a patient-defined 7-point Likert scale ranging from "substantially worse" to "substantially improved"
Global Improvement Scale (GIS) Scores Week 1 | Week 1
  The Global Improvement Scale is an overall assessment of Irritable Bowel Syndrome (IBS) symptoms using a patient-defined 7-point Likert scale ranging from "substantially worse" to "substantially improved"
Global Improvement Scale (GIS) Scores Week 4 | Week 4
  The Global Improvement Scale is an overall assessment of Irritable Bowel Syndrome (IBS) symptoms using a patient-defined 7-point Likert scale ranging from "substantially worse" to "substantially improved"
Global Improvement Scale (GIS) Scores Week 8 | Week 8
  The Global Improvement Scale is an overall assessment of Irritable Bowel Syndrome (IBS) symptoms using a patient-defined 7-point Likert scale ranging from "substantially worse" to "substantially improved"
Global Improvement Scale (GIS) Scores Week 12 | Week 12
  The Global Improvement Scale is an overall assessment of Irritable Bowel Syndrome (IBS) symptoms using a patient-defined 7-point Likert scale ranging from "substantially worse" to "substantially improved"

SECONDARY OUTCOMES:
Change in Perceived Stress Level (PSS) Scores | Baseline, Week 1, Week 4, Week 8, and Week 12
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress
Change in Five Factor Mindfulness Questionnaire (5FMQ) Scores | Baseline, Week 4, Week 8, and Week 12
  39-question measure that assesses trait mindfulness. In addition to the total score, there are five subscales: Non-judgement, Non-reaction, Describe, Observe, and Act with Awareness - Average scores are calculated by summing the responses and dividing by the number of items, and indicate the average level of agreement with the each subscale (1 = rarely true, 5 = always true). Higher scores are indicative of someone who is more mindful in their everyday life
Change in Mindful Eating Questionnaire (MEQ) Scores | Baseline, Week 8, and week 12
  28-question measure that assesses eating habits and mental tendencies while eating - Scoring. Each item was scored from 1 to 4, where higher scores signified more mindful eating. Each subscale score was calculated as the mean of items, excluding those with a "not-applicable" response. The summary score was the mean of the 5 subscales
Change in Positive and Negative Affect Schedule (PANAS_State) Questionnaire Scores | Baseline, Week 8, and Week 12
  20-question measure that assesses the degree to which positive and negative emotions are currently being felt - Positive Affect Score: Add the scores on items 1, 3, 5, 9, 10, 12, 14, 16, 17, and 19. Scores can range from 10 - 50, with higher scores representing higher levels of positive affect - Mean Scores: 33.3 (SD±7.2) Negative Affect Score: Add the scores on items 2, 4, 6, 7, 8, 11, 13, 15, 18, and 20. Scores can range from 10 - 50, with lower scores representing lower levels of negative affect - Mean Score: 17.4 (SD ± 6.2)
Change in cortisol blood levels | Baseline and Week 8
  differences in cortisol levels
Change in cytokine blood levels | Baseline and Week 8
  differences in cytokine levels - cytokine levels drawn at 8 am at screening or baseline if patient agrees - The detection of intracellular cytokines is a relatively new technique in which cells are permeabilized and antibodies are used to detect cytokine protein within cells by flow cytometry - when too many cytokines are released, it can cause your immune system to go into overdrive
Change in serotonin blood levels | Baseline and Week 8
  differences in serotonin levels
Change in Irritable Bowel Syndrome Quality of Life (IBS-QOL) Scores | Baseline, Week 4, Week 8, and Week 12
  The individual responses to the 34 items are summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS specific quality of life.
Change in Hospital Anxiety and Depression Scale (HADS) Scores | Baseline, Week 1, Week 4, Week 8, and Week 12
  The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression
Change in Irritable bowel syndrome symptom severity (IBS-SSS) Scores | Baseline, Week 1, Week 4, Week 8, and Week 12
  IBS-SSS is a composite score of abdominal pain, number of days with abdominal pain, bloating/distension, satisfaction with bowel habits, and IBS-related quality of life (QoL). Each measure is rated from 0 to 100, with total scores ranging from 0 to 500 - Mild, moderate and severe cases were indicated by scores of 75 to 175, 175 to 300 and > 300
Gastroparesis Cardinal Symptom Index (GCSI) Scores | Baseline, Week 1, Week 4, Week 8, and Week 12
  The GCSI total score is constructed as the average of the three symptom subscales. GCSI total score can range from 0 to 5, with higher scores reflecting greater symptom severity

CONTACTS AND LOCATIONS:
Overall Officials: Baharak Moshiree, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Gastroenterology and Hepatology Morehead Medical Plaza, Charlotte, North Carolina, United States